CLINICAL TRIAL: NCT03126214
Title: Improving Stroke Prevention in Atrial Fibrillation Through Pharmacist Prescribing: Program for the Identification of 'Actionable' AF (PIAAF) Rx Study
Brief Title: Improving Stroke Prevention in Atrial Fibrillation Through Pharmacist Prescribing
Acronym: PIAAFRx
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Canadian Stroke Prevention Intervention Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0024466
Record Dates: First submitted 2017-04-12; First posted 2017-04-24 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: atrial fibrillation; stroke; oral anticoagulation therapy; pharmacist case management
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Anticoagulants; Warfarin

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, randomized, stepped wedge trial design. Participants will be randomized to "early" (day 0-90) versus "delayed" pharmacist intervention (starting day 90-180).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Pharmacist Arm (Experimental): OAC therapy will be initiated/adjusted by the community pharmacist in accordance to the Canadian Cardiovascular Society Guidelines for the Management of Atrial Fibrillation.
  Interventions: Drug: Anticoagulants
- Enhanced Usual Care Arm (Active Comparator): Pharmacist will be refer participants to their physician in regards to OAC therapy for atrial fibrillation. The pharmacist will provide a current medication list to the physician as well as notification of a new diagnosis of atrial fibrillation
  Interventions: Drug: Anticoagulants

INTERVENTIONS:
Drug: Anticoagulants — Anticoagulant therapy will be initiated/titrated in patients with atrial fibrillation in accordance with the Canadian Cardiovascular Society Guidelines for Atrial Fibrillation.
  Other Names: warfarin and novel oral anticoagulants

SUMMARY:
The purpose of this study is to compare the effectiveness of prescribing oral anticoagulation therapy by pharmacist intervention compared to enhanced usual care in participants with unrecognized AF and/or known AF but not taking blood thinners.

DETAILED DESCRIPTION:
Background:

AF is the most common arrhythmia and the leading cause of stroke. Despite robust evidence oral anticoagulation (OAC) therapy is effective and safe for stroke prevention in patients with AF; there is a lack of real-world application. Alternative strategies to deliver stroke prevention therapy need to be explored. Although pharmacists' prescribing of antihypertensive and lipid lowering drug therapy has been shown to increase adherence to guideline-based targets and warfarin management improve control of international normalized ratios in anticoagulation clinics, the role of pharmacist initiation of OAC therapy compared to usual care in AF patients for stroke prevention in a community setting is unclear.

In this study, the investigators will screen participants presenting to community pharmacies to identify participants with unrecognized AF and/or known AF but not taking blood thinners or not on optimal OAC therapy and randomize care to either the pharmacist or enhanced usual care (family physician notification by pharmacist).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years with one additional stroke risk factor (hypertension, diabetes, heart failure history of or left ventricular ejection fraction <0.40), previous stroke or transient ischemic attack).
* Atrial fibrillation and not on oral anticoagulation (OAC) therapy but eligible
* Atrial fibrillation on sub-optimal OAC

Exclusion Criteria:

* Uncontrolled hypertension (defined as average SBP ≥ 160 mmHg [2 readings taken at time of screening]).
* End stage renal disease (CrCl < 15 ml/min)
* Valvular Heart Disease including those with prosthetic valve, mitral stenosis (moderate to severe) or valve repair.
* Excess alcohol intake (males: ≥ 28 units/week, females: ≥ 21 units/week. One unit of alcohol = 8 oz beer, 1 oz hard liquor or 4 oz wine).
* Intracranial bleed at any point.
* History of "Major Bleeding" at any point (defined as overt bleeding at a critical site including intracranial, intraspinal, intraocular, pericardial, or retroperitoneal; or bleed requiring hospitalization).
* Foreshortened life-expectancy or severe comorbidities precluding study follow-up period
* Unable to read/understand English
* Severe cognitive impairment (defined as score ≥ 5 on the Short Portable Mental Status Questionnaire)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Optimal Oral Anticoagulant (OAC) Therapy for Atrial Fibrillation Stroke Prevention | 3 months
  Proportion of participants receiving optimal OAC therapy in accordance with the Canadian Cardiovascular Society Guidelines for Atrial Fibrillation in the early intervention arm compared to the delayed intervention arm. Optimal defined as a new prescription for OAC in a previously untreated AF or known AF who should be on an OAC or adjustment of an existing OAC prescription.

SECONDARY OUTCOMES:
Prevalence of AF | Through study completion, an average of 1 year
  To determine the prevalence of participants with unrecognized AF eligible for OAC therapy and those with AF who should be on OAC therapy but are either not on or their existing OAC prescriptions; require adjustment due to contraindications, or sub-optimal levels (hereafter referred to those with "actionable" AF)
Patient Satisfaction with Pharmacists Services | 3 months
  Assessed using the validated Participant Satisfaction with Pharmacists Services Questionnaire (consists of 22 questions with 4 point Likert scale).
Qualitative Assessment of Implementation by Pharmacist | Through study completion, an average of 1 year
  Assessed using the questionnaire developed by the SEARCH-AF study
Healthcare Utilization | One year
  To determine the number of hospital, emergency department and physician visits related to AF
Healthcare Utilization | One year
  To determine the number of laboratory testing performed related to oral anticoagulation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Roopinder Sandhu, MD, MPH, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandhu RK, Fradette M, Lin M, Youngson E, Lau D, Bungard TJ, Tsuyuki RT, Dolovich L, Healey JS, McAlister FA. Stroke Risk Reduction in Atrial Fibrillation Through Pharmacist Prescribing: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2421993. doi: 10.1001/jamanetworkopen.2024.21993. PMID 39046741